CLINICAL TRIAL: NCT05793879
Title: Anomias Rehabilitation Training Through 360° Videos
Brief Title: Virtual Reality Training for Aphasia Rehabilitation
Acronym: Aphasia360
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Fondazione Poliambulanza (Unknown)
Responsible Party: Principal Investigator, Claudia Repetto, Associate Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC
Record Dates: First submitted 2023-03-07; First posted 2023-03-31 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Anomic Aphasia
Keywords: virtual reality; embodied cognition; rehabilitation
MeSH Terms: conditions — Anomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video 360 (Experimental): Patients will watch spherical videos displaying everyday actions towards objects; an audio is embedded describing the action and the object represented (i.e. "I'm cutting the potatoes").
  Interventions: Behavioral: Video 360
- Standard video (Active Comparator): Patients will watch standard videos displaying everyday actions towards objects; an audio is embedded describing the action and the object represented (i.e. "I'm cutting the potatoes")
  Interventions: Behavioral: Standard videos

INTERVENTIONS:
Behavioral: Video 360 — Patients will undergo 12 sessions, 3 per weeks, 4 weeks
  Arms: Video 360
Behavioral: Standard videos — Patients will undergo 12 sessions, 3 per weeks, 4 weeks
  Arms: Standard video

SUMMARY:
Aphasia is an acquired deficit following acute damage to the central nervous system that involves the difficulty or impossibility of understanding and formulating language. A typical disorder of non-fluent forms of aphasia is anomia. Anomia refers to the difficulty in finding words, in particular when trying to name objects and actions. According to the Embodied Cognition approach (EC), language is tightly connected to the motor system. In this view, language rehabilitation programs should stimulate language through the activation of the motor system. In this approach, since anomic deficits are often due to a weak link between the meaning of the word and its lemma, the Hebbs' principles of coincident and correlated learning can be exploited, i.e., by intensifying the synchronous activation of lexicon and semantics and connecting them with the motor counterpart. In this study, the investigators present an innovative training, based on the EC framework, in which they will make use of new technologies for anomia rehabilitation in post-stroke patients. Specifically, the researchers will use immersive 360° videos representing everyday actions displayed from the first-person point of view, experienced through a head-mounted display. The training will be administered 3 times a week for 4 weeks. The control group will watch standard videos representing the same actions recorded from the third-person perspective. Naming abilities will be tested before and after the training together with other cognitive and psychological measures. The investigators expect that the group who will undergo the 360° video-based training will show greater improvement of performance compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* naming disorder in the post-acute phase (index event occurring at least 6 months earlier)
* to have already received rehabilitation treatment in the acute phase
* noun naming below cut-off
* verbs naming below cut- off

Exclusion Criteria:

* concomitant or pre-existing (with respect to the index event) neurological and psychiatric deficits
* epilepsy
* balance disorders
* neglect

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of verbs and objects correctly named | post treatment, 1 month
  All the trained videos will be presented and the patient will be asked to name the verb and the object depicted. The accuracy will be registered

SECONDARY OUTCOMES:
Batteria per l'Analisi dei Deficit Afasici (BADA), naming subtest | post treatment, 1 month
  It is an Italian validated neuropsychological battery aiming at testing all the language abilities. It includes several tests tapping into the different linguistic abilities, but for the purpose of the present study only the verb and object naming subtest will be administered. Higher scores indicate greater naming abilities
EuroQol Health-related quality of life (EQ-5D-3L) | post treatment, 1 month
  The test consists of 2 sections. The first one is made of 5 questions scored from 1 to 5 points each. The final score ranges from 5 to 15, where the lesser the better. The second section is a visual scale on which the best state the patient can imagine is marked 100 and the worst state is marked 0.
Functional Outcome Questionnaire (FOQ-A) | post treatment, 1 month
  The survey is administered to the caregiver. It includes 32 questions each scored from 1 to 5 points. The final scores ranges from 32 to 160, where higher scores indicate greater communication abilities

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Repetto, Prof, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Poliambulanza, Brescia, Italy